CLINICAL TRIAL: NCT02161601
Title: Effect of Incorrectly Applied Cricoid Pressure During Rapid Sequence Induction. Evaluation With High-resolution Manometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Richard Pellrud, MD, Örebro University, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RAPESO-01; 2012/464 (Other: Regional Ethics Committe)
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Cricoid Pressure
Keywords: Cricoid pressure; Rapid Sequence Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Correctly and incorrectly applied cricoid pressure (Experimental)
  Interventions: Procedure: Cricoid Pressure

INTERVENTIONS:
Procedure: Cricoid Pressure — Correct Cricoid pressure applied against the cricoid cartilage, Incorrect Cricoid pressure applied against the thyroid cartilage and trachea

SUMMARY:
During emergency anesthesia (rapid sequence induction) , a firm pressure is applied to the cricoid cartilage of the patient in order to prevent passive regurgitation of gastric content into the pharynx. This maneuver is called cricoid pressure.

Cricoid pressure is often performed incorrectly, due to difficulties to locate the cricoid cartilage in many patients. Despite this, the effectiveness of an incorrectly applied cricoid pressure has not been investigated. In this study we have used high-resolution manometry (HRM) to evaluate pressures in the upper esophagus during correctly applied cricoid pressure (against the cricoid cartilage) compared to incorrectly applied cricoid pressure (against the thyroid cartilage and against the trachea) during a rapid sequence induction.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery and Anesthesia with intubation,
* ASA physical status I-II (American Society of Anesthesiologist classification system = system for assessing the fitness of cases before surgery)
* Body Mass Index > 18,5 and < 30
* Informed, signed and dated consent

Exclusion Criteria:

* Suspected difficult airway,
* Pharyngoesophageal dysfunction,
* Body Mass Index < 18,5 or > 30,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
difference in pressure (mmHg), detected by high resolution solid state manometry, between correctly vs incorrectly applied cricoid pressure | 15 sec. during ongoing cricoid pressure application

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University Hospital, Örebro, Sweden